CLINICAL TRIAL: NCT07083791
Title: AI-ECG Accessory Pathway Localisation Study
Acronym: AAPLS
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 347921
Record Dates: First submitted 2025-07-09; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Accessory Pathway; Artifical Intelligence; ECG
Keywords: AI-ECG; AI; ECG; Accessory pathway; Accessory pathway localisation
MeSH Terms: conditions — Pre-Excitation Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with manifest pre-excitation: Patients with a previous ECG demonstrating manifest pre-excitation, referred for an electrophysiology study as part of their clinical care

SUMMARY:
This study seeks to validate the real-world accuracy of an AI-based algorithm for identifying the location of an accessory pathway from the 12-lead electrocardiogram

DETAILED DESCRIPTION:
Silent validation study of an AI-ECG (artificial intelligence applied to electrocardiography) accessory pathway localisation algorithm, applied to prospective and consecutive cases in clinical practice, to determine its true accuracy and performance.

A pre-existing AI-ECG algorithm will be applied to participant ECG data, collected at the time of their clinical electrophysiology study (EPS) for ablation of their accessory pathway. This will be compared to the ground truth of the successful ablation location, determined by fluoroscopy and/or 3D electroanatomical mapping from their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Referred for EPS procedure as part of their clinical care, with a finding of pre-excitation on their ECG
* Manifest pre-excitation on their ECG any time prior to their procedure
* Able to give consent
* Minimum age 13 years old
* Maximum age 100 years old

Exclusion Criteria:

* Unable to give consent
* Adults > 100 years old
* Children < 13 years old
* Patients with known location of their accessory pathway from a previous EP study

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for an electrophysiology study +/- ablation, with evidence of previous pre-excitation on their 12-lead ECG.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Performance and accuracy of the AI-ECG accessory pathway localisation algorithm | At completion of recruitment, anticipated at 18 months
  Performance metrics of the AI-ECG accessory pathway localisation algorithm, including accuracy, F1-score, sensitivity, specificity, positive and negative predictive values. Benchmarked against the ground truth of human operator assessment from fluoroscopy and/or 3D electroanatomical mapping.

SECONDARY OUTCOMES:
Relative performance of the AI-ECG algorithm compared to human estimation | At completion of recruitment, anticipated at 18 months
  Difference in performance/accuracy between the AI-ECG accessory pathway localisation algorithm and human estimation from the 12-lead ECG
Relative performance of the AI-ECG algorithm compared to manual localisation algorithms | At completion of recruitment, anticipated at 18 months
  Difference in performance/accuracy between the AI algorithm and pre-specified, established manual localisation algorithms (Arruda, Milstein, Pambrun, Boersma, D'Avila and Chiang)
Accuracy of the ground truth locations from the human operator compared to the successful ablation location | At completion of recruitment, anticipated at 18 months
  The ground truth of successful ablation location determined by operator assessment of fluoroscopy ± 3D mapping will be compared to the true ablation location on a complete 3D electroanatomical annular map

CONTACTS AND LOCATIONS:
Overall Officials: Ahran Arnold, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT07083791/Prot_000.pdf
  • Informed Consent Form (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT07083791/ICF_001.pdf